CLINICAL TRIAL: NCT05940766
Title: Swiss 2024 Fever Monitoring Study: An Double-blinded, Randomized Controlled Multiple Crossover Superiority Trial on Continuous Fever Monitoring in Paediatric Patients With Cancer at Risk for Fever in Neutropenia
Brief Title: Swiss 2024 Continous Fever Monitoring in Pediatric Oncology Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Collaborators: ETH Zurich (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Supportive Care
Other Study IDs: Swiss 2024 Fever Monitoring
Record Dates: First submitted 2023-06-08; First posted 2023-07-11 (Actual); Last update posted 2023-07-11 (Actual); Status verified 2023-07

CONDITIONS: Pediatric Oncology Patients With Risk for Infections
Keywords: Fever; Neutropenia; Pediatric oncology; Core temperature; Wearable device; Continous monitoring; Automated alerts
MeSH Terms: conditions — Fever; Neutropenia

STUDY DESIGN:
Intervention Model Description: Prospective interventional, multi-center, double-blinded, randomized controlled, multiple crossover superiority trial
Who Masked: Participant, Investigator
Masking Description: Double-blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention "With CFM alerts" arm (Experimental): * Routine clinical care, which includes, among others, discrete fever measurements using ear thermometers in case of clinical deterioration or suspected fever, at the discretion of patients where applicable, parents and the treating team
  * Plus CFM with a CORE® WD running, with alerts being sent automatically to participants if the CFM detects an estimated core body temperature fulfilling the fever criterion of the respective study site (≥38.5°C or 39.0°C).
  Interventions: Other: Automated fever alerts
- Control "Without CFM alerts" arm (No Intervention): * Routine clinical care as in "With CFM alerts"
  * Plus CFM with a CORE® WD running as in "With CFM alerts", but with alerts being sent only if a clinically dangerous temperature of ≥40.0°C is detected, which will very rarely be the case before fever is detected by routine clinical care.

INTERVENTIONS:
Other: Automated fever alerts — Fever alerts are automated sent to participants if fever is detected
  Arms: Intervention "With CFM alerts" arm

SUMMARY:
In children and adolescents undergoing chemotherapy for cancer, fever in neutropenia (FN) is the most frequent potentially lethal complication of chemotherapy for cancer. Emergency hospitalization and empirical treatment with i.v. broad-spectrum antibiotics have reduced lethality from >50% in certain high risk situations to <1%. Fever without neutropenia is a further complication requiring emergency evaluation and often emergency treatment.

Continuous monitoring of fever leads to earlier fever detection compared to the usual discrete fever measurements performed only for clinical reasons. Earlier detection of fever leads to earlier assessment and treatment and thus can reduce the risk of complications.

This study primarily aims to assess, in pediatric patients undergoing chemotherapy for cancer, the efficacy of automated fever alerts resulting from continuous fever monitoring (CFM) using a wearable device (WD), measured by the duration of intravenous antibiotics (i.v. AB) given for any cause.

DETAILED DESCRIPTION:
Primary objective

The primary objective of this study is to determine if CFM fever alerts (CFM-FA) automatically sent by a WD reduce the duration of i.v. antibiotics application in children and adolescents treated with myelosuppressive chemotherapy for cancer.

Secondary objectives

Regarding safety

A. Number of fever episodes (FE) with safety relevant events (SREs)

B. Number of false alerts

C. Number of missed alarms

Regarding efficacy

D. Delay of chemotherapy application

E. Duration of antimicrobial application except i.v. antibiotics

F. Number of FEs diagnosed below or at temperature limit (TL) versus above TL

G. FEs according to chemotherapy intensity

H. WD measured core temperature at time of fever detection by ear thermometer

I. FEs reported outside TARs

J. Quality of life Questionnaire

K. Assessment of the side-effects of the WD

Tertiary objective

L. Comparison of continuously recorded core temperature of the WD with results of discrete measurements of tympanic temperature

M. Pattern search using data mining

ELIGIBILITY:
Inclusion Criteria:

* Chemotherapy treatment because of any malignancy expected to last ≥2 months at time of recruitment for myelosuppressive therapy, or at least 1 cycle of myeloablative chemotherapy followed by hematopoietic stem cell transplantation
* Age ≥1 month and <18 years at time of recruitment
* Written informed consent from patients and/or parents

Exclusion Criteria:

* Neonates <1 months
* Local skin disease prohibiting wearing of the WD
* Denied written informed consent from patients and/or parents
* Inclusion of vulnerable participants mandatory as vital signs and FN episodes differ significantly in children and adults

Ages: 1 Month to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 250 (Estimated)
Dates: Start 2024-10-01 (Estimated); Primary Completion 2028-05-31 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
The primary objective of this study is to determine if CFM fever alerts (CFM-FA) automatically sent by a WD reduce the duration of i.v. antibiotics application in children and adolescents treated with myelosuppressive chemotherapy for cancer. | 3 to 9 month per patient
  The cumulative duration of i.v. antibiotics applied

SECONDARY OUTCOMES:
Number of fever episodes (FE) with safety relevant events (SREs) | 3 to 9 month per patient
  Number of FE with SREs
Number of false alerts | 3 to 9 month per patient
  Number of false alerts
Number of missed alarms | 3 to 9 month per patient
  Number of missed alarms
Delay of chemotherapy application | 3 to 9 month per patient
  Duration of delay of chemotherapy application in days
Duration of antimicrobial application except i.v. antibiotics | 3 to 9 month per patient
  Duration of antimicrobial application except i.v. antibiotics
Number of fever episodes (FE) diagnosed below or at temperature limit (TL) versus above TL | 3 to 9 month per patient
  Number of FEs diagnosed below or at TL versus above TL
FEs according to chemotherapy intensity | 3 to 9 month per patient
  Amount of fever episodes according to chemotherapy intensity
Wearable Device (WD) measured core temperature at time of fever detection by ear thermometer | 3 to 9 month per patient
  WD measured core temperature at time of fever detection by ear thermometer
FEs reported outside times of risk (TARs) | 3 to 9 month per patient
  Amount of fever episodes reported outside TARs
Quality of life Questionnaire | Month 1, 6 and at study completion, an average of 1 year
  Proportion of participants indicating that wearing a WDs is acceptable/unacceptable, not increasing anxiety/increasing anxiety, providing/not providing security, increase burden/effort or not
Assessment of the side-effects of the WD | Through study completion, an average of 1 year
  Side effects reported by participants, if applicable

OTHER OUTCOMES:
Comparison of continuously recorded core temperature of the WD with results of discrete measurements of tympanic temperature | Through study completion, an average of 1 year
  Difference between discrete measurements of core temperature
Vital sign pattern search in monitored core temperature using data mining | Through study completion, an average of 1 year
  Exploration of potential changes in or specific patterns of all measured temperature signals within 48 hours before clinical diagnosis of fever

CONTACTS AND LOCATIONS:
Overall Officials: Eva K Brack, MD, PhD, Principal Investigator — Childrens' Clinic Bern, Inselspital, Bern
Locations (1):
- Childrens' Clinc Bern, Inselspital Bern, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: Yes
Publication in international journal of study protocol and results
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: End of study
Access Criteria: All study information will be made publically available as long as the patient as signed the informed consent for data sharing